CLINICAL TRIAL: NCT01194310
Title: Longtime Efficiency of Combined Cataract-Surgery and Excimer-Laser-Trabeculotomy or Trabectome in Glaucoma Surgery
Brief Title: Phaco vs. Phaco-ELT vs. Phaco-Trabectome 12m
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Phako/ELT/Trabectome-12m
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Glaucoma; Cataract
Keywords: glaucoma; cataract
MeSH Terms: conditions — Glaucoma; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- phaco alone: patients w/ diagnosis of open angle glaucoma underwent phaco alone
  Interventions: Procedure: phaco
- phaco-ELT: patients w/ diagnosis of open angle glaucoma underwent combined phaco plus ELT
  Interventions: Procedure: phaco; Procedure: phaco-ELT
- phaco-Trabectome: patients w/ diagnosis of open angle glaucoma underwent combined phaco plus Trabectome
  Interventions: Procedure: phaco; Procedure: phaco-Trabectome

INTERVENTIONS:
Procedure: phaco — Standard clear cornea phacoemulsification plsu intraocular lens Implantation (phaco) alone
Procedure: phaco-ELT — Standard clear cornea phacoemulsification plsu intraocular lens Implantation (phaco) plus excimer laser trabeculotomy (ELT)
  Groups: phaco-ELT
Procedure: phaco-Trabectome — Standard clear cornea phacoemulsification plsu intraocular lens Implantation (phaco) plus Trabectome
  Groups: phaco-Trabectome

SUMMARY:
This study compares efficacy (i.e. IOP and hypotensive medications) of phaco alone vs. combined phaco plus excimer laser trabeculotomy vs. combined phaco plus trabectome.

DETAILED DESCRIPTION:
Glaucoma is one of the most common reasons for blindness. Usually an elevated drain resistance is the reason, while aqueous humor production is normal. Medical reduction of intraocular pressure (IOP) is first line therapy in most cases. The gold standard of surgical treatment still is trabeculectomy (TE) but TE has a lot of drawbacks. In particular when glaucoma and cataract coexists, the investigators therefore prefer the combined procedure cataract extraction plus excimer laser trabeculotomy (ELT) or plus Trabectome. Indication is cataract and a moderate elevated IOP without medical therapy or a moderate cataract and elevated IOP with medical therapy.

The ELT is performed by an AIDA XeCl-Excimer Laser System (TUI-Laser AG, Germering, 1,2 mJ per burst, burst duration 16 ns, wave length 308 nm, spot diameter 200 µm). 10 foramina were made over 90 degrees of the anterior chamber angle. Trabectome procedure is performed with the Trabectome unit from Neomedix.

* Trial with medical device
* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria:

* All patients, which had Phaco, Phako/ELT, or Phaco-Trabectome from 01/2008 until 12/2011, where screened 12 month after surgery

Exclusion criteria:

* IOP >35 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toteberg-Harms M, Hanson JV, Funk J. Cataract surgery combined with excimer laser trabeculotomy to lower intraocular pressure: effectiveness dependent on preoperative IOP. BMC Ophthalmol. 2013 Jun 24;13:24. doi: 10.1186/1471-2415-13-24. PMID 23799932